CLINICAL TRIAL: NCT04304638
Title: Real-world Treatment Patterns and Clinical Outcomes in Epidermal Growth Factor Receptor(EGFR)-Mutant Unresectable Locally Advanced NSCLC: A Retrospective Multi-center Study
Brief Title: Real-world Treatment Patterns and Clinical Outcomes in EGFR-mutant Unresectable Locally Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Luhua Wang, Principal Investigator, Clinical Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CAMS19/216-2000
Record Dates: First submitted 2020-03-05; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Non Small Cell Lung Cancer; Stage III Non-small-cell Lung Cancer; EGFR Mutation-Related Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Radiation(Chemo-radiation): Patients in this group had been treated with definitive radiation/Chemo-radiation followed by no treatment until progression.
  Interventions: Radiation: radiation or chemo-radiation
- radiation+EGFR-TKI: Patients in this group had been treated with one of the following three ways: 1) definitive radiation and concurrent EGFR-TKI followed by EGFR-TKI till progression; 2) EGFR-TKI followed by radiation and continue TKI util progression; 3) radiation and TKI thereafter until progression.
  Interventions: Radiation: radiation or chemo-radiation; Drug: EGFR-TKI Inhibitor
- EGFR-TKI: Patients in this group had been treated with EGFR-TKI without any other treatment until progression.
  Interventions: Drug: EGFR-TKI Inhibitor

INTERVENTIONS:
Radiation: radiation or chemo-radiation — standard treatment for stage III lung cancer
  Groups: Radiation(Chemo-radiation); radiation+EGFR-TKI
Drug: EGFR-TKI Inhibitor — the standard treatment for stage IV lung cancer with EGFR mutation
  Other Names: EGFR-TKI alone
  Groups: EGFR-TKI; radiation+EGFR-TKI

SUMMARY:
The investigators will obtain a cohort of patients from multiple large cancer centers in China and try to unravel the efficacy of "radiotherapy combined with EGFR-TKI", which may provide some evidences for the treatment of stage III-inoperable NSCLC.

DETAILED DESCRIPTION:
The frequency of EGFR mutations in patients with stage III inoperable adenocarcinoma or non-squamous cell carcinoma is 17-31%, which is relatively low. Compared to patients with EGFR wild type, the efficacy of radiotherapy or chemo-radiotherapy may be different in EGFR mutant patients. Some small sample studies showed, compared with patients with EGFR wild type, patients with EGFR mutations have a lower risk of local recurrence and a higher risk of distant metastasis under the standard treatment for stage III lung cancer, which demonstrate the strength of systemic therapy may help. Radiotherapy combined with EGFR-Tyrosine kinase inhibitors(TKI) is a feasible treatment strategy. In view of the low mutation frequency and few prospective research results, the investigators try to explore the survival differences of three treatment strategies used in clinical practice based on the real world data. The investigators will obtain a cohort of patients from multiple large cancer centers in China and try to unravel the efficacy of "radiotherapy combined with EGFR-TKI", which may provide some evidences for the further study.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed NSCLC with adenocarcinoma
* stage III (AJCC 7th edition)
* inoperable or refuse surgery
* EGFR-TKI mutation, specimen from tissue or blood

Exclusion Criteria:

* the pathology was not adenocarcinoma
* stage I,II and IV
* anaplastic lymphoma kinase (ALK) rearrangement
* no follow-up data achievable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stage III patients with EGFR mutation.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
median progression-free survival (mPFS) | Tumor scans had been performed at baseline, and every 3 months after the first treatment of EGFR-TKI or the last dose of radiation (whichever occurs first) in 5 years
  The time of half patients who are alive and progression-free after the disease diagnose, estimated by the Kaplan-Maier method and using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
median overall survival(mOS) | Tumor scans had been performed at baseline, and every 3 months after the first treatment of EGFR-TKI or the last dose of radiation (whichever occurs first) in 5 years
  The time of half patients who are alive after the disease diagnose, estimated by the Kaplan-Maier method and using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
failure pattern | Tumor scans had been performed at baseline, and every 3 months after the first treatment of EGFR-TKI or the last dose of radiation(whichever occurs first) in 5 years
  Rate of disease failure in local, regional and distant sites.

CONTACTS AND LOCATIONS:
Overall Officials: Luhua Wang, MD, Principal Investigator — Cancer center of Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No